CLINICAL TRIAL: NCT05470075
Title: A Multicenter, Randomized, Double-blind, Dose Finding, Parallel Controlled With Active Drug and Placebo, Phase II Clinical Trial to Evaluate the Efficacy and Safety of HR18042 Tablets for Postoperative Analgesia After Impacted Teeth Removal Surgery
Brief Title: A Study to Evaluate the Efficacy and Safety of HR18042 Tablets for Postoperative Analgesia After Impacted Teeth Removal Surgery.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor's R&D strategy is adjusted.
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR18042-202
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, double-blind, dose finding, parallel controlled with active drug and placebo, phase II clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Experimental A: HR18042 175mg (Experimental)
  Interventions: Drug: HR18042 tablets
- Experimental B: HR18042 225mg (Experimental)
  Interventions: Drug: HR18042 tablets
- Experimental C: HR18042 275mg (Experimental)
  Interventions: Drug: HR18042 tablets
- Active Drug Comparator：Tramadol hydrochloride SR Tablets 100mg (Active Comparator)
  Interventions: Drug: Tramadol hydrochloride SR Tablets
- Placebo Comparator: Placebos match to HR18042 and Tramadol hydrochloride SR Tablets (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: HR18042 tablets — Drug: HR 18042 tablets 175mg and placebos match to Tramadol hydrochloride SR Tablets Dosing frequency: single dose; Route of administration: oral
  Arms: Experimental A: HR18042 175mg
Drug: HR18042 tablets — Drug: HR 18042 tablets 225mg and placebos match to Tramadol hydrochloride SR Tablets Dosing frequency: single dose; Route of administration: oral
  Arms: Experimental B: HR18042 225mg
Drug: HR18042 tablets — Drug: HR 18042 tablets 275mg and placebos match to Tramadol hydrochloride SR Tablets Dosing frequency: single dose; Route of administration: oral
  Arms: Experimental C: HR18042 275mg
Drug: Tramadol hydrochloride SR Tablets — Drug: Tramadol hydrochloride SR Tablets 100mg and placebos match to HR18042 tablets Dosing frequency: single dose; Route of administration: oral
  Arms: Active Drug Comparator：Tramadol hydrochloride SR Tablets 100mg
Drug: Placebos — Drug: Placebos match to HR18042 tablets and Tramadol hydrochloride SR Tablets Dosing frequency: single dose; Route of administration: oral
  Arms: Placebo Comparator: Placebos match to HR18042 and Tramadol hydrochloride SR Tablets

SUMMARY:
This is a multicenter, randomized, double-blind, dose finding, parallel controlled with active drug and placebo, phase II clinical trial, and the purpose of the study is to evaluate the efficacy and safety of HR18042 tablets for postoperative analgesia after impacted teeth removal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Scheduled to remove the impacted tooth.
3. Any NRS score reaches the inclusion criteria within 4 hours after the surgery.
4. Willing to comply with the study procedures and requirements.
5. Willing and able to provide written informed consent for this study.

Exclusion Criteria:

1. Subjects who have used other drugs that have the analgesic effect.
2. Subjects who have used any drug that affect the efficacy and safety of study drug.
3. Subjects who have infection or other complications on the planned oral surgical site.
4. Subjects with hypertension or hypotension during screening period.
5. Subjects with severe cardiovascular and cerebrovascular diseases.
6. Subjects with severe gastrointestinal disease.
7. Subjects with Respiratory diseases.
8. Subjects with a history of seizure, or drug or alcohol abuse.
9. Subjects with significant abnormal electrocardiogram result.
10. Subjects with significant abnormal laboratory value.
11. Subject who were allergic to the study drug and ingredients.
12. Pregnancy, lactation or having recent pregnant plan.
13. Subjects who participated in other clinical research study 30 days before entering this study.
14. Other conditions unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
the Sum of Pain Intensity Differences (SPID) using numerical rating scale (NRS, ranging from 0-10, the larger the number, the more severe the pain) within 4 hours after drug administration | 0-4 hours after drug administration

SECONDARY OUTCOMES:
the Sum of Pain Intensity Differences (SPID) using numerical rating scale (NRS, ranging from 0-10, the larger the number, the more severe the pain) within 6 hours, 8 hours and 12 hours after drug administration | 0 - 6 hours, 8 hours and 12 hours after drug administration
the Differences of Pain Intensity (PID) from each evaluating timepoint to baseline using numerical rating scale (NRS, ranging from 0-10, the larger the number, the more severe the pain) after drug administration | 0-12 hours after drug administration
Pain relief degree at each evaluating timepoint using pain relief scale (PAR, ranging from 0-4, the larger the number, the more obvious the pain relief) after drug administration | 0-12 hours after drug administration
Sum of pain relief degree using pain relief scale (PAR, ranging from 0-4, the larger the number, the more obvious the pain relief) within 4 hours, 6 hours, 8 hours, 12 hours after drug administration (SPAR) | 0 - 4 hours, 6 hours, 8 hours and 12 hours after drug administration
Proportion of subjects who reach a 50% reduction in pain intensity from baseline using numerical rating scale (NRS, ranging from 0-10, the larger the number, the more severe the pain) at each evaluating timepoint | 0-12 hours after drug administration
Time from drug administration to the first NRS score≤3 | 0-12 hours after drug administration
Time from drug administration to the first use of rescue medication | 0-12 hours after drug administration
Proportion of subjects who receive rescue therapy during the treatment period | 0-12 hours after drug administration]
Subject's overall satisfaction score of the study medication using subject satisfaction scale (ranging from 0-10, the larger the number, the higher the satisfaction) | 12 hours after drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Stomatology Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided